CLINICAL TRIAL: NCT05861128
Title: An Open-Label, Multicenter, Extension Study to Assess the Long-Term Safety and Efficacy of Jaktinib in Patients With Active Ankylosing Spondylitis(AS)
Brief Title: Extension Study to Evaluate Safety and Efficacy of Jaktinib in Patients With Active Ankylosing Spondylitis(AS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK030
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jaktinib 100mg BID (twice daily) (Experimental)
  Interventions: Drug: Jaktinib

INTERVENTIONS:
Drug: Jaktinib — Participants will receive 100 mg Jaktinib orally twice daily for 32 weeks

SUMMARY:
The purpose of this study is to determine if Jaktinib is safe and effective in participants with active ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* The investigators concluded that the participants continued to benefit from treatment with Jaktinib.
* The participants have been fully informed and voluntarily signed informed consent.
* The participants completed the ZGJAK029 study for 16 weeks of treatment and visitation and had good compliance.
* The interval between the participants' first dose and the last dose of ZGJAK029 ≤ 4 weeks.

Exclusion Criteria:

* There were any grade ≥3 adverse events within 4 weeks prior to enrollment and no return to grade 1 or normal.
* Within 4 weeks prior to enrollment, participants had the following infectious diseases: tuberculosis infection requiring treatment; HIV-positive, syphilis, HBV infection, HCV infection.
* The investigators considered participants unsuitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Related Discontinuations at 32 Weeks | Baseline up to Week 32
  Treatment-emergent AEs were events that occurred between first dose of study drug and up to 32 weeks that were absent before treatment or that worsened relative to pretreatment state.

SECONDARY OUTCOMES:
Percentage of Participants Achieving ASAS20 Response at Week 4, 8, 12, 16，20，24，28 and 32 | Baseline, Week 4, 8, 12, 16，20，24，28 and 32
  ASAS20 assess 4 domains: PGA of Disease (assess disease activity on a scale of 0 [not active] to 10 [very active], high score=more disease activity), total back pain (scale of 0 [no pain] to 10 [most severe pain], high score=more severity), Function (BASFI; participant's level of ability on scale of 0 [easy] to 10 [impossible], low score= better functional health) and Inflammation (morning stiffness, Mean of Q5 and Q6 of BASDAI defined as 6-item questionnaire measure disease activity on a scale of 0 [none] to 10 [severe], high score=more disease activity). ASAS20 response: >= 20% improvement from baseline in disease activity and absolute change of >=1 unit in >=3 domains and no worsening of >=20% and an absolute change of >=1 unit in remaining domain.
Percentage of Participants Achieving ASAS40 Response at Week 4, 8, 12, 16，20，24，28 and 32 | Baseline, Week 4, 8, 12, 16，20，24，28 and 32
  ASAS40 assessed 4 domains: the "PGA" (assess disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity), total back pain (on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (from BASFI: assess participant's level of ability on a scale of 0 [easy] to 10 [impossible], lower scores= better functional health) and Inflammation (morning stiffness, Mean of Q5 and Q6 of BASDAI defined as 6 item questionnaire: measures disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity). ASAS40 response: >=40% and >=2 units improvement in >=3 domains and no worsening at all in the remaining domain.
Change From Baseline in Patient's Assessment of Spinal Pain: Total Back Pain at Week 4, 8, 12, 16，20，24，28 and 32 | Baseline, Week 4, 8, 12, 16，20，24，28 and 32
  Participants marked their level of total back pain on a numerical rating scale (NRS) ranged from 0 (no pain) to 10 (most severe pain), with higher scores indicated more severe pain.
Percentage of Participants Achieving ASAS 5/6 Response at Week 4, 8, 12, 16，20，24，28 and 32 | Baseline, Week 4, 8, 12, 16，20，24，28 and 32
  ASAS 5/6 consists of 6 domains: 4 used in ASAS20 - PGA (assess disease activity on a scale of 0 [not active] to 10 [very active], higher score=more disease activity), Spinal Pain (total back pain) (on a scale of 0 [no pain] to 10 [most severe pain], higher score=more severity), Function (using BASFI which assess participant's level of ability on a scale of 0 [easy] to 10 [impossible], lower scores= better functional health) and Inflammation (using BASDAI, mean of Q 5 and 6, which assess disease activity on a scale of 0 [none] to 10 [severe], higher score=more disease activity), CRP (was measured in mg per liter) and Spinal mobility was measured in centimeter and calculated as mean of right and left measurements of lateral spinal flexion from BASMI. ASAS 5/6: defined as >=20% improvement in at least 5 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China